CLINICAL TRIAL: NCT01936272
Title: Neurocognitive Outcomes and Changes in Brain and Cerebral Spinal Fluid (CSF) Volume After Treatment of Post-Infectious Hydrocephalus (PIH) in Ugandan Infants by Shunting Versus ETV/CPC
Brief Title: Randomized Controlled Trial of Shunt vs ETV/CPC for PIH in Ugandan Infants
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Boston Children's Hospital (Other)
Collaborators: Penn State University (Other); The Hospital for Sick Children (Other); CURE Children's Hospital, Uganda (Other)
Responsible Party: Principal Investigator, Benjamin C. Warf, Professor of Neurosurgery, Hydrocephalus and Spina Bifida Chair, Boston Children's Hospital
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: P00002785
Record Dates: First submitted 2013-07-29; First posted 2013-09-06 (Estimated); Last update posted 2023-08-16 (Actual); Status verified 2023-08

CONDITIONS: Hydrocephalus
MeSH Terms: conditions — Hydrocephalus

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Chhabra Shunt Placement (Active Comparator): The shunting arm will comprise a standard frontal approach ventriculoperitoneal shunt using a silastic Chhabra system.
  Interventions: Device: Chhabra Shunt Placement
- ETV/CPC (Active Comparator): The Endoscopic Third Ventriculostomy/Choroid Plexus Cauterization (ETV/CPC) arm will comprise a standard frontal approach with flexible endoscopy.
  Interventions: Procedure: ETV/CPC

INTERVENTIONS:
Device: Chhabra Shunt Placement
  Arms: Chhabra Shunt Placement
Procedure: ETV/CPC
  Arms: ETV/CPC

SUMMARY:
Two treatment options exist for infant patients with hydrocephalus. Most patients are treated with a surgical procedure in which a shunt is inserted into the brain and abdomen. In recent years, however, another treatment has developed called Endoscopic Third Ventriculostomy (ETV) with Choroid Plexus Cauterization (ETV/CPC).This research study is being done to measure the results of these procedures in children less than six months of age who have hydrocephalus as the result of a brain infection, called post-infectious hydrocephalus, or PIH. This study will evaluate patients in more detail to measure brain growth and development.

DETAILED DESCRIPTION:
World over, infants with hydrocephalus are mainly treated using a shunt, which is a device made of soft plastic tubing that moves extra fluid from the brain to the abdomen. Surgery is required to insert a shunt into the brain and the abdomen. In recent years, we have developed another treatment called Endoscopic Third Ventriculostomy (ETV) with Choroid Plexus Cauterization (ETV/CPC). This research study is being done to measure the results of these procedures in children less than six months of age who have hydrocephalus as the result of a brain infection, called post-infectious hydrocephalus, or PIH. This is the most common cause of hydrocephalus in Ugandan babies. This study will evaluate patients in more detail to measure brain growth and development. Children in the study will have special testing to measure developmental progress as well as special imaging to evaluate the progress of their brain growth.

ELIGIBILITY:
Inclusion Criteria:

* Infants less than 180 days (six months) old
* Symptomatic hydrocephalus
* Post-infectious Hydrocephalus based on clinical and CT parameters2
* Must be from the following Ugandan districts: Bugiri, Busia, Iganga, Jinja, Kampala, Kamuli, Kapchorwa, Katakwi, Kumi, Mayuge, Mbale, Mukono, Pallisa, Sironko, Soroti, and Tororo

Exclusion Criteria:

* Any patient with a scalp erosion or infection that would exclude the patient from shunt implantation
* Any patient with ventricular loculations that would normally indicate the use of ventriculoscopy as an adjunct to shunt placement
* Any patient with absence of any visible cortical mantle on the CT
* Patients must be appropriate candidates for either surgical procedure - shunt placement alone or ETV/CPC

Ages: 1 Day to 180 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2013-05-27 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change of Age-normed Bayley Scales of Infant Development (BSID)-III scores | 12 months and 24 months post treatment
  Neurocognition will be measured using the BSID-III Cognitive Scale. Change will be assessed at 24 months post treatment from baseline score (12 months post treatment).

SECONDARY OUTCOMES:
Brain Volume | 12 months, 24 months, 5 years, and 7-10 years post treatment
  Volume unit of measure is cubic millimeters. Volume is measured using CT scans.
CSF Volume | 12 months, 24 months, 5 years, and 7-10 years post treatment
  Volume unit of measure is cubic millimeters. Volume is measured using CT scans.
Vineland Adaptive Behavior Scales | 5 years and 7-10 years post treatment
  The primary purpose of the VABS is to assess the social abilities of school age children.

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin C Warf, MD, Principal Investigator — Boston Children's Hospital
Locations (1):
- CURE Children's Hospital Uganda, Mbale, Uganda

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared with researchers outside of the study team.

REFERENCES:
- [Derived] Harper JR, Cherukuri V, O'Reilly T, Yu M, Mbabazi-Kabachelor E, Mulando R, Sheth KN, Webb AG, Warf BC, Kulkarni AV, Monga V, Schiff SJ. Assessing the utility of low resolution brain imaging: treatment of infant hydrocephalus. Neuroimage Clin. 2021;32:102896. doi: 10.1016/j.nicl.2021.102896. Epub 2021 Nov 23. PMID 34911199
- [Derived] Punchak M, Mbabazi Kabachelor E, Ogwal M, Nalule E, Nalwoga J, Ssenyonga P, Mugamba J, Rattani A, Dewan MC, Kulkarni AV, Schiff SJ, Warf B. The Incidence of Postoperative Seizures Following Treatment of Postinfectious Hydrocephalus in Ugandan Infants: A Post Hoc Comparison of Endoscopic Treatment vs Shunt Placement in a Randomized Controlled Trial. Neurosurgery. 2019 Oct 1;85(4):E714-E721. doi: 10.1093/neuros/nyz122. PMID 31086941
- [Derived] Kulkarni AV, Schiff SJ, Mbabazi-Kabachelor E, Mugamba J, Ssenyonga P, Donnelly R, Levenbach J, Monga V, Peterson M, MacDonald M, Cherukuri V, Warf BC. Endoscopic Treatment versus Shunting for Infant Hydrocephalus in Uganda. N Engl J Med. 2017 Dec 21;377(25):2456-2464. doi: 10.1056/NEJMoa1707568. PMID 29262276